CLINICAL TRIAL: NCT07355296
Title: PODOMOUNT-Basket, a Phase II, Multicentre, Randomised, 2-arm Parallel-group, Double-blind, Placebo-controlled Basket Trial to Assess Safety, Tolerability, PK, and Efficacy of BI 764198 in Four Proteinuric Kidney Diseases
Brief Title: PODOMOUNT-Basket, a Study to Test Whether BI 764198 Helps Adults and Adolescents With Different Types of Kidney Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1434-0027; 2025-523425-17 (Registry Identifier: CTIS); U1111-1328-7108 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2026-01-20; First posted 2026-01-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Proteinuric Kidney Diseases

STUDY DESIGN:
Intervention Model Description: basket trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Secondary focal segmental glomerulosclerosis (sFSGS) cohort (Experimental)
  Interventions: Drug: BI 764198
- Treatment resistant primary Minimal Change Disease (TR-pMCD) cohort (Experimental)
  Interventions: Drug: BI 764198
- Alport Syndrome cohort (Experimental)
  Interventions: Drug: BI 764198
- Treatment resistant primary Membranous Nephropathy (TR-pMN) cohort (Experimental)
  Interventions: Drug: BI 764198
- Placebo cohort (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 764198

INTERVENTIONS:
Drug: BI 764198 — BI 764198
  Arms: Alport Syndrome cohort; Secondary focal segmental glomerulosclerosis (sFSGS) cohort; Treatment resistant primary Membranous Nephropathy (TR-pMN) cohort; Treatment resistant primary Minimal Change Disease (TR-pMCD) cohort
Drug: Placebo matching BI 764198 — Placebo matching BI 764198
  Arms: Placebo cohort

SUMMARY:
This study is open to adults with certain kidney conditions, including secondary focal segmental glomerulosclerosis (sFSGS), treatment-resistant primary minimal change disease (TR-pMCD), Alport Syndrome (AS), and treatment-resistant primary membranous nephropathy (TR-pMN). Adolescents with treatment-resistant primary MCD can also participate in this study. The purpose of this study is to find out whether a medicine called BI 764198 helps people with these kidney conditions.

Participants are put into 2 groups randomly, which means by chance. One group takes BI 764198 tablets, and the other group takes placebo tablets. Placebo tablets look like BI 764198 tablets but do not contain any medicine. Participants take a tablet once a day for 20 weeks. All participants also continue their standard medication for their kidney condition during the study. Participants have twice the chance of being placed in the BI 764198 group than in the placebo group.

Participants are in the study for about 7 months. During this time, they visit the study site 6 times and have 3 phone calls. Doctors regularly test the protein levels in participants' urine by collecting urine samples. They also check kidney function by taking blood samples. The results are compared between the two groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years of age (≥12 years of age for Treatment resistant primary Minimal Change Disease (TR-pMCD)) on the day of signing informed consent/assent (Visit 1)
* Body Mass Index (BMI) of ≤40 kg/m2 at screening visit (Visit 1)
* Weight of ≥40 kg at screening
* Estimated glomerular filtration rate (eGFR) ≥25 mL/min/1.73 m2 (chronic kidney disease (CKD) EPI formula based on serum cystatin C) at screening visit

  * For adult participants (≥18); ≥25 mL/min/1.73 m2 (CKD-EPI formula based on serum cystatin C) at the screening visit
  * For adolescent participants (<18); ≥25 mL/min/1.73 m2 (chronic kidey disease under 25 years (CKiD U25) formula using height and serum cystatin C) at the screening visit
* Seated blood pressure (mean of 3 values) systolic blood pressure (SBP) ≤160 mmHg (adult participants ≥18) or SBP ≤140 mmHg (participants <18) at the screening visit (Visit 1). A participant with a documented history of white coat hypertension may be included as long as the participant is considered medically stable by the investigator and "true" blood pressure can be considered to be ≤160 mmHg (adult participants ≥18) or ≤140 mmHg (adolescent participants <18)
* Participants should be treated with angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs), at a stable optimised dose for at least 8 weeks prior to the screening visit (Visit 1), with no plan to change the dose until the end of the randomised treatment period (i.e. end of trial (EoT), Week 20) unless not tolerated or indicated as per the discretion of the investigator
* If treated with (non-steroidal) mineralocorticoid receptor antagonist (MRA), endothelin receptor antagonists (ERA), glucagon-like peptide-1 (GLP-1) or Sodium-glucose co-transporter-2 (SGLT2) inhibitors (SGLT2i), participants must be on a stable dose for at least 8 weeks prior to the screening visit (Visit 1), preferably with no plan to change the dose until the end of the randomised double-blind treatment period (i.e. EoT, Week 20)
* Participants treated with oral immunosuppressive therapy except glucocorticoids (e.g. Calcineurin inhibitor(s) (CNI), mycophenolate mofetil/-sodium, cyclophosphamide) must be on a stable dose for at least 12 weeks prior to the screening visit (Visit 1) with no plans to change their dose during the trial treatment period
* Patients treated/to be treated with oral glucocorticoids have to be at a dose ≤10 mg/d prednisolone or equivalent for ≥4 weeks prior to screening with no plan to increase the dose during the treatment period.

Further inclusion criteria apply.

Exclusion Criteria:

* A history of organ transplantation or planned transplantation during the course of the study
* Use of intravenous immunosuppressive agents (e.g. cyclophosphamide, rituximab, obinutuzumab) in the past 6 months prior to screening visit (Visit 1)
* Participants in whom initiation of oral or IV immunosuppression is anticipated during the course of the trial
* Treatment with metformin or dofetilide (multidrug and toxin extrusion protein 1 (MATE1) substrates) within one week prior to randomisation visit (Visit 2) through 5 days after the EoT visit
* Treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (CYP3A4/5) within one week or 5 half-lives (whichever is longer) prior to randomisation visit (Visit 2)
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >3X the upper limit of normal (ULN) at screening visit (Visit 1)
* Clinically significant laboratory abnormalities or medical conditions which pose a safety risk for the participant or may interfere with the trial objectives in the investigator's opinion (except for renal function tests or deviation of clinical laboratory values that are related to the podocytopathy in question) at screening visit
* QTc intervals (QTcF) greater than 450 ms in males or greater than 470 ms in females, or any other clinically relevant ECG findings (at the investigator's discretion) at screening visit (Visit 1) Further exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-12-24 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Relative change from baseline to Week 20 in 24-hr Urine protein-to-Creatinine Ratio (UPCR) | At baseline and week 20

SECONDARY OUTCOMES:
Treatment response, defined as at least 25% relative reduction in 24-hr UPCR from baseline to Week 20 | At baseline and week 20
Treatment response, defined as at least 40% relative reduction in 24-hr UPCR from baseline to Week 20 | At baseline and week 20
Absolute change in estimated glomerular filtration rate (eGFR) in mL/min/1.73m2 (based on cystatin C) from baseline to Week 20 | At baseline and week 20

CONTACTS AND LOCATIONS:
Locations (120):
- United States (18):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Amicis Research Center - Balboa, Granada Hills, California
  - Academic Medical Research Institute - Glendale, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Colorado Kidney Center, Denver, Colorado
  - Florida Kidney Physicians - Boca Raton, Boca Raton, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Panoramic Health, Riverview, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - New York Nephrology and Dialysis Access Surgery, PC, Clifton Park, New York
  - NYU Langone Nephrology Associates-Mineola, Mineola, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Provecta Researh Network, Houston, Texas
  - West Virginia University Medicine, Morgantown, West Virginia
- Argentina (2):
  - Clinica Privada Velez Sarfield, Córdoba
  - CardioAlem Investigaciones, San Isidro
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Belgium (4):
  - AZORG Ziekenhuis, Aalst
  - ULB Hopital Erasme, Brussels
  - Az Maria Middelares Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (4):
  - Universidade Federal do Ceará, Fortaleza
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Fundação Oswaldo Ramos (Hospital do Rim), São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo
- Canada (3):
  - CaRe Clinic (Calgary), Calgary, Alberta
  - Victoria Hospital (LHSC), London, Ontario
  - Maisonneuve-Rosemont Hospital, Monteral, Quebec
- China (12):
  - Peking University First Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The First People's Hospital of Nanning, Nanning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - People's Hospital of Sichuan Province, Sichuan
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen
- Croatia (5):
  - Specialty Hospital Medico, Rijeka
  - General Hospital Vinkovci, Vinkovci
  - Clinical Hospital Sveti Duh, Zagreb
  - Solmed Polyclinic, Zagreb
  - University Hospital Dubrava, Zagreb
- Zealand University Hospita; Roskilde, Roskilde, Denmark
- Tartu University Hospital, Tartu, Estonia
- France (5):
  - CHU Amiens-Picardie, Amiens
  - HOP Pellegrin, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - HOP Pasteur, Nice
  - Hôpital Necker, Paris
- Germany (5):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - General University Hospital of Patras, Pátrai
- India (4):
  - Aartham Multi Super Speciality Hospital, Ahmedabad
  - AIIMS Bhubaneshwar, Bhubaneshwar
  - Government Medical College, Kozhikode
  - Noble Hospital Pvt Ltd, Pune
- Italy (4):
  - Azienda Universitaria Ospedaliera Consorziale Policlinico Bari, Bari
  - Policlinico S. Orsola-Malpighi, Bologna
  - Asst Santi Paolo E Carlo, Milan
  - Fondazione Salvatore Maugeri, Pavia
- Japan (4):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Aichi, Nagoya
  - The Jikei University Hospital, Tokyo, Minato-ku
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
- Netherlands (3):
  - Amsterdam UMC Locatie AMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
- Norway (4):
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (5):
  - Central Clinical Hospital of the Medical University of Lodz, Lodz
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Pomorski Uniwersytet Medyczny w Szczecinie, Samodzielny Publiczny Szpital Kliniczny nr 2, Szczecin
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny Im. Jozefa Polikarpa Brudzinskiego W Warszawie, Warsaw
  - Central Clinical Hospital of the Ministry of National Defence - Military Institute of Medicine, Warsaw
- Portugal (5):
  - Unidade Local de Saúde de Almada-Seixal E.P.E., Almada
  - ULS Braga, Braga
  - ULS de São José, Lisbon
  - Unidade Local de Saúde Lisboa Occidental, E.P.E, Lisbon
  - ULS de Loures-Odivelas, E.P.E, Loures
- Romania (2):
  - Institutul Clinic Fundeni, Bucharest
  - County Emergency Hospital "Pius Brinzeu" Timisoara, Timișoara
- Slovakia (3):
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - FMC Dialysis Services Kosice, Košice
  - Univ. Hospital Martin, Martin
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (3):
  - Danderyds Sjukhus, Danderyd
  - Universitetssjukhuset, Linköping, Linköping
  - Uppsala University Hospital, Uppsala
- Klinik Hirslanden, Zurich, Switzerland
- Taiwan (4):
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (6):
  - Adana City Hospital, Adana
  - Ankara Etlik City Hospital, Ankara
  - Bursa Uludag University, Bursa
  - İstanbul Çapa University, Istanbul
  - Kocaeli University Faculty of Medicine Hospital, İzmit
  - Erciyes University, Melikgazi/Kayseri
- United Kingdom (4):
  - Bradford Institute for Health Research, Bradford
  - The Royal London Hospital, London
  - King's College Hospital, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency